CLINICAL TRIAL: NCT03075657
Title: Study of add-on Ramelteon Therapy on Sleep and Circadian Rhythm Disruption in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T/IM-NF/Pharma/01/17
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; ramelteon; Haloperidol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The rating of PANSS and PSQI will be done by one Psychiatrist who will be blind to the groups and treatment alloted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Risperidone group (Active Comparator): Schizophrenia patients with predominant negative symptoms on Risperidone monotherapy
  Interventions: Drug: Risperidone
- Risperidone with Ramelteon group (Experimental): Schizophrenia patients with predominant negative symptoms on Risperidone with add-on Ramelteon therapy
  Interventions: Drug: Risperidone and Ramelteon
- Haloperidol group (Active Comparator): Schizophrenia patients with predominant positive symptoms on Haloperidol monotherapy
  Interventions: Drug: Haloperidol
- Haloperidol with Ramelteon group (Experimental): Schizophrenia patients with predominant positive symptoms on Haloperidol with add-on Ramelteon therapy
  Interventions: Drug: Haloperidol and Ramelteon

INTERVENTIONS:
Drug: Risperidone — Risperidone will be prescribed at dose of 2 mg per day
  Arms: Risperidone group
Drug: Risperidone and Ramelteon — Ramelteon will be prescribed 8mg/day as an add-on therapy to Risperidone 2 mg per day
  Arms: Risperidone with Ramelteon group
Drug: Haloperidol — Haloperidol will be prescribed at a dose of 4 mg per day
  Arms: Haloperidol group
Drug: Haloperidol and Ramelteon — Ramelteon will be prescribed 8mg/day as an add-on therapy to Haloperidol 4 mg per day
  Arms: Haloperidol with Ramelteon group

SUMMARY:
The proposed study has been planned to evaluate the effect of add-on ramelteon on sleep pattern/quality and circadian rhythm disruption in patients with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a mental dysfunction of thought, perception and behaviour which can be attributed to complex and dynamically interacting perturbations in multiple neurochemical systems. Along with these cardinal features of schizophrenia, sleep disorders and disturbed circadian rhythm are commonly encountered among patients. Markedly decreased sleep efficiency, delayed sleep onset and frequent awakenings are most common observations. Endogenous melatonin is a dependable biomarker of circadian rhythmicity and, it has already been found that the nocturnal rise of endogenous melatonin is blunted leading to circadian dysrhythmia in schizophrenia.

The antipsychotics prescribed for the condition though cause improvement in the cardinal symptoms of the disease but have no significant effect on melatonin levels. The blunted peak of night time melatonin secretion are not restored or even decreased even after several months therapy with antipsychotics. In this clinical scenario, add-on therapy with sedative/ hypnotics along with antipsychotics is mandate for a prescription. Previous studies revealed that add-on therapy with benzodiazepines can worsen the already existing derangement in circadian rhythm by decreasing secretion of nocturnal melatonin. A long term add on therapy with benzodiazepines in patients on antipsychotics has been found to have an increased risk of death.

Addition of melatonin to the pharmacotherapy of schizophrenia elevates mood and daytime functioning in addition to improved sleep in schizophrenia patients. Melatonin, apart from being a hypnotic and circadian rhythm restoring compound, also possess neuroprotective, anti-neuroinflammatory and antioxidant properties. The rate limiting step of melatonin biosynthetic pathway is the alkylation of serotonin to N- acetyl serotonin, catalyzed by enzyme AANAT (aryl-alkylamine- N-acetyl-transferase). Study of AANAT enzyme and its modulation to achieve normal rhythmical secretion of melatonin can also be a potential target for resynchronising the circadian rhythm.

Ramelteon is a melatonin receptor agonist approved for treatment of insomnia by the USFDA. It exerts its action by acting on MT1 and MT2 receptors at suprachiasmatic nucleus. The long term safety of ramelteon has been evaluated by several workers and found no significant adverse effects like abuse liability, rebound insomnia and cognitive impairment. In contrast to melatonin, it shows higher-binding affinity for MT1 and MT2 receptors, more lipophilic and has a longer half-life(t1/2 of melatonin is 20-50 min whereas that of ramelteon is 1-2.6 hrs and that of its active melabolite M-II is 2-5 hrs). In addition, ramelteon has been already evaluated as a potential adjunctive treatment for learning and memory deficits in schizophrenia.

The sleep and circadian rhythm disorders in schizophrenia have so far been given very less importance by researchers and there are limited studies targeting or modulating the melatonin pathway. Therefore, proposed study has been planned to evaluate the effect of add-on ramelteon on sleep pattern/quality and circadian rhythm disruption in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients of either sex with age range 18-65 years with the clinical diagnosis of schizophrenia. (DSM-V)
* Treatment naïve patients or patients who had not taken any treatment for at least 4 weeks before inclusion.
* Legal guardian of patients consenting to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Schizoaffective disorder or schizophrenia with somatoform disorders.
* Highly agitated patients who need immediate treatment.
* Patients who are already under treatment for the presenting conditions.
* Patients with comorbid substance abuse or history of organicity
* Patients with known history of dementia, obstructive sleep apnoea syndrome, diabetes mellitus.
* Pregnant and nursing women.
* History of allergy or hypersensitivity to ramelteon.
* Legal guardian of patients not willing to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in serum melatonin over 4 weeks from baseline | Baseline and 4 weeks
  ELISA

SECONDARY OUTCOMES:
Change in quality of sleep over 4 weeks from baseline | Baseline and 4 weeks
  Pittsburgh Sleep Quality Index (PSQI) scoring
Change in urinary melatonin(6MTs) over 4 weeks from baseline | Baseline and 4 weeks
  HPLC
Change in serum AANAT enzyme over 4 weeks from baseline | Baseline and 4 weeks
  ELISA
Change in severity of symptoms of schizophrenia over 4 weeks from baseline | Baseline and 4 weeks
  PANSS Scoring

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, DM, Study Chair — AIIMS, BHUBANESWAR
Locations (1):
- All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohrs S. Sleep disturbances in patients with schizophrenia : impact and effect of antipsychotics. CNS Drugs. 2008;22(11):939-62. doi: 10.2165/00023210-200822110-00004. PMID 18840034
- [Result] Wehr TA, Aeschbach D, Duncan WC Jr. Evidence for a biological dawn and dusk in the human circadian timing system. J Physiol. 2001 Sep 15;535(Pt 3):937-51. doi: 10.1111/j.1469-7793.2001.t01-1-00937.x. PMID 11559786
- [Result] Afonso P, Figueira ML, Paiva T. Sleep-promoting action of the endogenous melatonin in schizophrenia compared to healthy controls. Int J Psychiatry Clin Pract. 2011 Nov;15(4):311-5. doi: 10.3109/13651501.2011.605954. Epub 2011 Aug 28. PMID 22122006
- [Result] Wulff K, Dijk DJ, Middleton B, Foster RG, Joyce EM. Sleep and circadian rhythm disruption in schizophrenia. Br J Psychiatry. 2012 Apr;200(4):308-16. doi: 10.1192/bjp.bp.111.096321. Epub 2011 Dec 22. PMID 22194182
- [Result] Mann K, Rossbach W, Muller MJ, Muller-Siecheneder F, Pott T, Linde I, Dittmann RW, Hiemke C. Nocturnal hormone profiles in patients with schizophrenia treated with olanzapine. Psychoneuroendocrinology. 2006 Feb;31(2):256-64. doi: 10.1016/j.psyneuen.2005.08.005. Epub 2005 Sep 26. PMID 16185814
- [Result] Cohrs S, Pohlmann K, Guan Z, Jordan W, Meier A, Huether G, Ruther E, Rodenbeck A. Quetiapine reduces nocturnal urinary cortisol excretion in healthy subjects. Psychopharmacology (Berl). 2004 Jul;174(3):414-20. doi: 10.1007/s00213-003-1766-6. Epub 2004 Jan 20. PMID 14735295
- [Result] Robinson S, Rosca P, Durst R, Shai U, Ghinea C, Schmidt U, Nir I. Serum melatonin levels in schizophrenic and schizoaffective hospitalized patients. Acta Psychiatr Scand. 1991 Sep;84(3):221-4. doi: 10.1111/j.1600-0447.1991.tb03133.x. PMID 1950621
- [Result] Monteleone P, Natale M, La Rocca A, Maj M. Decreased nocturnal secretion of melatonin in drug-free schizophrenics: no change after subchronic treatment with antipsychotics. Neuropsychobiology. 1997;36(4):159-63. doi: 10.1159/000119377. PMID 9396013
- [Result] Hajak G, Rodenbeck A, Bandelow B, Friedrichs S, Huether G, Ruther E. Nocturnal plasma melatonin levels after flunitrazepam administration in healthy subjects. Eur Neuropsychopharmacol. 1996 May;6(2):149-53. doi: 10.1016/0924-977x(96)00005-3. PMID 8791041
- [Result] Kabuto M, Namura I, Saitoh Y. Nocturnal enhancement of plasma melatonin could be suppressed by benzodiazepines in humans. Endocrinol Jpn. 1986 Jun;33(3):405-14. doi: 10.1507/endocrj1954.33.405. PMID 3757924
- [Result] Baandrup L, Fagerlund B, Jennum P, Lublin H, Hansen JL, Winkel P, Gluud C, Oranje B, Glenthoj BY. Prolonged-release melatonin versus placebo for benzodiazepine discontinuation in patients with schizophrenia: a randomized clinical trial - the SMART trial protocol. BMC Psychiatry. 2011 Oct 5;11:160. doi: 10.1186/1471-244X-11-160. PMID 21975110
- [Result] Lavie P. Melatonin: role in gating nocturnal rise in sleep propensity. J Biol Rhythms. 1997 Dec;12(6):657-65. doi: 10.1177/074873049701200622. PMID 9406042
- [Result] Suresh Kumar PN, Andrade C, Bhakta SG, Singh NM. Melatonin in schizophrenic outpatients with insomnia: a double-blind, placebo-controlled study. J Clin Psychiatry. 2007 Feb;68(2):237-41. doi: 10.4088/jcp.v68n0208. PMID 17335321
- [Result] Miyamoto M. Pharmacology of ramelteon, a selective MT1/MT2 receptor agonist: a novel therapeutic drug for sleep disorders. CNS Neurosci Ther. 2009 Winter;15(1):32-51. doi: 10.1111/j.1755-5949.2008.00066.x. PMID 19228178
- [Result] Johnson MW, Suess PE, Griffiths RR. Ramelteon: a novel hypnotic lacking abuse liability and sedative adverse effects. Arch Gen Psychiatry. 2006 Oct;63(10):1149-57. doi: 10.1001/archpsyc.63.10.1149. PMID 17015817
- [Result] Spadoni G, Bedini A, Lucarini S, Mor M, Rivara S. Pharmacokinetic and pharmacodynamic evaluation of ramelteon : an insomnia therapy. Expert Opin Drug Metab Toxicol. 2015 Jul;11(7):1145-56. doi: 10.1517/17425255.2015.1045487. Epub 2015 May 8. PMID 25956235
- [Result] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771